CLINICAL TRIAL: NCT04750486
Title: Lower Limb Compression Prevents Hypotension After Epidural in Labor: A Randomized Controlled Trial
Brief Title: Lower Limb Compression Prevents Hypotension After Epidural in Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Laura Mroue, MD, Principal Investigator, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB# 20-07-2555
Record Dates: First submitted 2021-01-29; First posted 2021-02-11 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Labor Pain; Maternal Hypotension
Keywords: Epidural anesthesia; Lower extremity compression
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: Randomization of patients to either control or study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (No Intervention): No intervention, the patient will be provided routine care at time of epidural placement without use of sequential compression devices.
- Lower Extremity Compression (Experimental): Patients will have sequential compression devices prior to epidural placement, and maintained for at least one hour following procedure.
  Interventions: Device: Sequential compression devices

INTERVENTIONS:
Device: Sequential compression devices — Two lower limb intermittent compression devices to be placed on the mid-calf of each leg.
  Other Names: Lower extremity intermittent compression devices
  Arms: Lower Extremity Compression

SUMMARY:
The goal of this study is to determine whether the use of sequential compression devices (lower limb compression) can reduce the rate of maternal hypotension after epidural, and therefore reduce the incidence of fetal heart tracing complications during labor.

DETAILED DESCRIPTION:
Maternal hypotension during epidural anesthesia in laboring patients can cause a number of problems for both mother and fetus. Despite standard anesthesia protocols designed to minimize the occurrence of hypotension during epidural placement, approximately 30% of laboring patients will still experience clinically significant hypotension. Maternal hypotension can affect placental blood flow causing fetal bradycardia and academia, as well as maternal symptoms such as dizziness, nausea, and vomiting. Therefore, there is a need for improved management of women in labor at time of epidural placement to avoid negative consequences for mother and fetus. We plan to investigate whether the use of lower limb compression devices at the time of epidural would decrease maternal hypotension.

Pregnant women who request epidural anesthesia during labor will be recruited and enrolled in this single site, randomized controlled trial. Patients will be randomized into either control or sequential compression device (SCD) groups. Following epidural, blood pressures will be measured at 1, 5, 15, 30, 45, and 60 minutes and rates of hypotension with subsequent fetal heart tracing abnormalities will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Women with pregnancy at term (greater than or equal to 37 weeks 0 days gestation)
* Singleton gestation
* In labor (spontaneous or induced)
* Requested epidural for pain management

Exclusion Criteria:

* Any diagnosis of hypertension or cardiovascular disease
* Any contraindications to lower extremity compression including deep venous thrombosis in past 6 months, infected leg wound, or deformity of lower extremity
* Any contraindications to epidural placement including severe thrombocytopenia and spinal deformity

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Maternal hypotension | Blood pressures measured at 1 minute following epidural placement.
  Determined by maternal blood pressure measurements.
Maternal hypotension | Blood pressures measured at 5 minutes following epidural placement.
  Determined by maternal blood pressure measurements.
Maternal hypotension | Blood pressures measured at 15 minutes following epidural placement.
  Determined by maternal blood pressure measurements.
Maternal hypotension | Blood pressures measured at 30 minutes following epidural placement.
  Determined by maternal blood pressure measurements.
Maternal hypotension | Blood pressures measured at 45 minutes following epidural placement.
  Determined by maternal blood pressure measurements.
Maternal hypotension | Blood pressures measured at 60 minutes following epidural placement.
  Determined by maternal blood pressure measurements.

SECONDARY OUTCOMES:
Fetal heart rate tracing category | Two hours following epidural placement.
  Determination of category I, II or III fetal heart rate tracing.
Delivery method | length of labor.
  Vaginal or cesarean delivery ( report)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Johnson, MD, Study Director — Detroit Medical Center/Wayne State University
Locations (1):
- Detroit Medical Center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brizgys RV, Dailey PA, Shnider SM, Kotelko DM, Levinson G. The incidence and neonatal effects of maternal hypotension during epidural anesthesia for cesarean section. Anesthesiology. 1987 Nov;67(5):782-6. doi: 10.1097/00000542-198711000-00025. No abstract available. PMID 3674479
- [Background] Goetzl LM; ACOG Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin. Clinical Management Guidelines for Obstetrician-Gynecologists Number 36, July 2002. Obstetric analgesia and anesthesia. Obstet Gynecol. 2002 Jul;100(1):177-91. doi: 10.1016/s0029-7844(02)02156-7. PMID 12100826
- [Background] Corke BC, Datta S, Ostheimer GW, Weiss JB, Alper MH. Spinal anaesthesia for Caesarean section. The influence of hypotension on neonatal outcome. Anaesthesia. 1982 Jun;37(6):658-62. doi: 10.1111/j.1365-2044.1982.tb01278.x. PMID 7091625
- [Background] American Society of Anesthesiologists Task Force on Obstetric Anesthesia. Practice guidelines for obstetric anesthesia: an updated report by the American Society of Anesthesiologists Task Force on Obstetric Anesthesia. Anesthesiology. 2007 Apr;106(4):843-63. doi: 10.1097/01.anes.0000264744.63275.10. No abstract available. PMID 17413923